CLINICAL TRIAL: NCT04266938
Title: Impact of Rapid ART Initiation on Retention in Care in the Southern US
Acronym: RAPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Bailey Benidir, PharmD, Clinical Pharmacist, University of Louisville
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 20.0017
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prospective RAPID (Active Comparator): The prospective RAPID arm will include all patients who meet inclusion criteria and who start BIC/F/TAF within 7 days of HIV diagnos
  Interventions: Behavioral: Rapid start of antiretrovirals
- Prospective Non- RAPID (Active Comparator): The prospective non-RAPID arm will include all patients identified as having new HIV diagnosis per health department records, but who failed to establish care at the 550 Clinic and begin BIC/F/TAF within one week of diagnosis
  Interventions: Behavioral: Non- RAPID start
- Retrospective Non- RAPID (Active Comparator): The retrospective Non-RAPID arm will include historic controls who enrolled in the treatment program from 2012, when universal ART guidelines were implemented, until prior to the implementation of RAPID start of ART.
  Interventions: Behavioral: Retrospective analysis

INTERVENTIONS:
Behavioral: Rapid start of antiretrovirals — Utilize health navigators to link patients with newly diagnosed HIV into care and treatment within 7 days
  Arms: Prospective RAPID
Behavioral: Retrospective analysis — Review historical standard of care relative to time to start antiretrovirals and impact on retention in care.
  Arms: Retrospective Non- RAPID
Behavioral: Non- RAPID start — Review of patients who failed to establish care and start ART within 7 days of HIV diagnosis and analyze impact on retention in care.
  Arms: Prospective Non- RAPID

SUMMARY:
Impact of Rapid ART Initiation on Retention in Care in the Southern US

Specific Goals and Aims:

The major goal for this study is to determine if rapid start of antiretroviral (ART) therapy increases retention in HIV medical care. The investigators hypothesize that there will be an increase in retention in care with rapid start, by removing barriers that would normally delay enrollment in a treatment program and enforce the importance of linkage to care and ART initiation from diagnosis.

In order to test this hypothesis, the investigators have the following specific aims for their proposed study:

1. Study retention in care after rapid ART start in comparison to standard of care.
2. Analyze risk factors for decreased retention in care, with focus on high-risk populations.
3. Analyze potential demographic and geographic determinants of retention in care.
4. Generate retention in care data in a Southern US state.

The investigators hypothesize the introduction of rapid start ART, as well as the introduction of care navigators, will lead to improved clinical outcomes, including retention in care at one year, viral suppression at one year, time to viral suppression, and time to first missed appointment. In the event rapid start ART fails to have a positive impact on clinical outcomes, the results of this study will still positively contribute to the knowledge gap, since there is a scarcity of data in the Southern United States, specifically in high-risk populations, such as racial and ethnic minorities, youth, and patients co-infected with hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Prospective arms: Human subjects ≥18 years old, newly diagnosed with HIV who are establishing care at the 550 Clinic.
* Retrospective arm: Human subjects ≥18 years old, newly diagnosed with HIV who established care at the 550 Clinic and were treated with ART between 2012-2019.

Exclusion Criteria:

* Pregnancy
* Prior HIV diagnosis or exposure to ART
* Medical necessity for therapy with ART agent other than bictegravir/emtricitabine/tenofovir alafenamide (BIC/F/TAF), such as drug allergy, drug-drug interactions, creatinine clearance <30.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Retention in Care | 12 months
  Retention in HIV care at one year after initiation of rapid ART start, defined as 1) keeping at least 3 visits within the first 12 months of care and 2) attending a clinic visit between months 9-15 of the 12-month mark and 3) experiencing no gaps in care greater than 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- 550 Clinic, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No